CLINICAL TRIAL: NCT06746129
Title: Day 3 Versus Day 5 Embryo Transfer in IVF Patients With Few Embryos
Brief Title: Cleavage-stage Versus Blastocyst-stage Embryo Transfer in IVF Patients With Few Embryos
Acronym: PRECiSE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Brigham and Women's Hospital (Other); Boston IVF (Other); Columbia University (Other); Weill Medical College of Cornell University (Other); Mayo Clinic (Other); University of Michigan (Other); Patient-Centered Outcomes Research Institute (Other); Massachusetts General Hospital (MGH) (Unknown); Yale University (Other); UCSF Center for Reproductive Health (Unknown); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Werner Neuhausser, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024P000892; 35477 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2024-12-14; First posted 2024-12-24 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Infertility (IVF Patients)
Keywords: infertility; in vitro fertilization; cleavage stage embryo; blastocyst; embryo transfer
MeSH Terms: conditions — Infertility | interventions — Embryo Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cleavage-stage embryo transfer (Active Comparator): embryo(s) will be transferred on day 3 of embryo development (cleavage-stage embryo)
  Interventions: Procedure: embryo transfer
- blastocyst embryo transfer (Active Comparator): embryo(s) will be transferred on day 5-7 of embryo development (blastocyst-stage embryo)
  Interventions: Procedure: embryo transfer

INTERVENTIONS:
Procedure: embryo transfer — transfer of embryo(s) into the uterine cavity

SUMMARY:
Infertility affects more than 6 million women the United States and is a major life event that results in a wide range of socio-cultural, emotional, physical and financial problems. The most successful treatment for infertility, in-vitro fertilization (IVF), fertilizes a woman's eggs with her partner's sperm in a culture dish and transfers the resulting embryos into the uterus. Most of the time, prior to being transferred, embryos are grown in the dish for 5-7 days after which some of them reach an advanced stage (blastocyst stage). This has several advantages such as a lower chance of a multiple pregnancies (twins, triplets etc.) after transfer and fewer transfer procedures. However, it is possible that embryos would survive better if transferred into the uterus at the 8-cell stage after growing them for only 3 days. Thus, when patients only have a small number of embryos they and their physicians face the difficult choice when to transfer because there are currently no studies available to guide this decision.

This randomized controlled trial is comparing pregnancy outcomes and patient satisfaction of poor prognosis patients with 5 or fewer embryos undergoing either transfer of an advanced (blastocyst) or an 8-cell embryo.

This study will provide the data for the development of guidelines for IVF providers to make evidence-based decisions when to transfer embryos in poor prognosis IVF patients, reduce patients' anxiety regarding cycle cancellation and improve patient counseling, which will increase patients' ability to participate in the development of their treatment plan.

DETAILED DESCRIPTION:
Background and Significance:

It is a major unanswered question for many IVF patients and their providers whether embryos which did not develop into a blastocyst after in vitro culture to day 5-7 of development may have resulted in a pregnancy when transferred into the uterus on day 3, at the cleavage (8-cell) stage. For patients with few (<=5) embryos there is a lack of studies analyzing pregnancy outcomes with either type of embryo transfer (ET). As a result of this uncertainty, these patients and their providers face the difficult clinical decision when to transfer their embryos. This decision is often based on 'expert opinion' and driven by patient anxiety about embryo survival in vitro but not high-quality evidence. Thus, patients with few embryos often receive cleavage-stage transfers forgoing the advantages of blastocyst transfer such as the possibility to transfer a single embryo (SET) which reduces the incidence of multiple pregnancies without reducing the live birth rate per ET.

The investigators are working with nine IVF centers across the US to enroll 1126 patients age 18-44 who are treated for infertility with IVF for the first time and have 5 or fewer embryos. The investigators will assign an equal number of patients by chance to either the 8-cell embryo or the blastocyst transfer group. If there are any surplus embryos that meet freezing criteria they will be frozen and then thawed and transferred in a subsequent cycle. The investigators will monitor patients for 6 months or until all embryos are transferred and, if pregnancy is achieved, until delivery (9 months). For each group the investigators will measure the chance to have a live birth per cycle (primary outcome) and the risk of miscarriage, multiple pregnancy, cycle cancellation (secondary) outcomes based on clinical assessments.

The investigators are working with patients, advocacy groups (RESOLVE, Fertility within Reach), professional societies in reproductive medicine (ASRM, NEFS), clinicians, embryologists, nurses, implementation experts, and a health psychologist, as well as payer (Optum, Winfertility) and policymaker (ASRM, NEFS) representatives to design, and conduct this study and implement the results.

Study Aims:

The goal of the proposed research is to compare the cumulative life birth rate per egg retrieval and the risk of adverse pregnancy outcomes for cleavage-stage versus blastocyst ET in patients with few (<=5) embryos. The investigators hypothesize that blastocyst is superior to cleavage-stage ET in patients with ≤5 zygotes with regard to the primary outcome of cumulative live birth per oocyte retrieval and that there may be differences in other patient-relevant pregnancy outcomes between these two types of ET. Our long-term objective is to develop and implement evidence-based practice guidelines and patient counseling tools for the timing of ET in poor prognosis IVF patients.

Study Description:

This multicenter, randomized, controlled, parallel two-group 1:1 trial compares cleavage-stage vs. blastocyst ET in patients undergoing IVF treatment for infertility within a network of 9 academic IVF centers in the US. The study population consists of first autologous cycle IVF patients ages 18- 44 years with ≤5 zygotes on day 1 of embryo development. The investigators will enroll 563 participants per treatment arm, for a total sample size of 1126. The demographics of the study population at BIVF/BIDMC and other enrolling sites across the US represents that of women seeking care for infertility and reproductive disorders with a mean age of 36.3 years and a mean BMI of 27.4. The investigators expect 69% to be Caucasian, 5% African American, 10% Hispanic, 15% Asian, and 1% Pacific.

The investigators selected outcomes on the basis of importance to patients, providers and other stakeholders:

Primary: cumulative live birth rate per retrieval ('take home baby rate') Secondary: multiple live birth, miscarriage, cycle cancellation Exploratory: time to pregnancy, number of involved procedures, ectopic pregnancy, live birth rate/fresh ET, adverse perinatal outcomes (stillbirth, preterm birth), financial burden, patient satisfaction/psychological distress, facilitators and barriers for patient involvement in the timing of ETs and for implementation and adoption of uniform blastocyst transfer Pre-specified subgroup Analyses: Subgroups of interest are participants with age < 38y and ≥ 38y, <=2 versus 3-5 zygotes, from different ethnic subgroups and poor versus good quality cleavage-stage embryos undergoing single embryo transfer.

Patients will be followed for 6 months after the egg retrieval or until all embryos generated in the cycle have been transferred. All pregnancy outcomes will be assessed from the time of a positive pregnancy test to delivery (9months).

Analytic Methods:

The planned sample size of 1126 participants, equally distributed across the two intervention arms, will provide an estimated power of 99.4%, 91.2% and 80% for a 13.7%, 10% and 8.4% difference in CLBR, respectively. The investigators based our sample size calculation on a 0.05-level two-sided Fisher's exact test for a difference in proportions assuming a 10% cross-over and 10% loss to follow-up rate. Importantly, this sample size will also provide adequate power to determine differences in the secondary outcomes with 80% power.

Stakeholders:

The investigators are working with patients, advocacy groups (RESOLVE, Fertility within Reach), professional societies in reproductive medicine (ASRM, NEFS), clinicians, embryologists, nurses, implementation experts, and a health psychologist, as well as payer (Optum, Winfertility) and policymaker (ASRM, NEFS) representatives to design, and conduct this study and implement the results.

ELIGIBILITY:
Inclusion Criteria:

* First autologous IVF cycle
* ≤5 zygotes on day 1 of development
* Fresh embryo transfer

Exclusion Criteria:

* Planned preimplantation genetic testing (PGT)
* History of recurrent pregnancy loss (≥3)
* Body mass index >40
* Presence of uterine factor infertility
* Planned gestational carrier
* Endometrial lining <6mm measured on the day of trigger
* Lupron-only trigger, elevated progesterone in the fresh cycle (≥1.5ng/ml)
* Delayed fertilization (>18 hours)
* Rescue intracytoplasmic sperm injection (following failed regular fertilization)
* Use of non-ejaculated sperm (testicular sperm extraction)
* Embryo transfer number outside American Society of Reproductive Medicine (ASRM) guidelines
* Cycle is converted to a cycle in which all embryos are frozen

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1126 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
cumulative live birth per IVF cycle | month 9 after embryo transfer
  the number of live births resulting from transfer of all embryos obtained from one egg retrieval

SECONDARY OUTCOMES:
multiple pregnancy | month 9 after embryo transfer
  rate of twin, triplet and higher order pregnancies
number of involved procedures | month 9 after embryo transfer
  number of embryo transfers necessary to achieve pregnancy and procedures to treat pregnancy complications
ectopic pregnancy | month 9 after embryo transfer
  rate of pregnancies outside the uterus (Fallopian tube, cervix, ovary, abdomen)
live birth rate/fresh embryo transfer | month 9 after embryo transfer
  rate of birth of a live baby per embryo transfer performed
adverse perinatal outcomes (stillbirth, preterm birth) | month 9 after embryo transfer
  rate of pregnancy complications such as still birth, preterm birth, abruption etc
financial burden | month 9 after embryo transfer
  cost of treatment for cleavage stage and blastocyst embryo transfer
Incidence of patient satisfaction/psychological distress | month 9 after embryo transfer
  The investigators will use a mixed method approach with a satisfaction questionnaire in combination with semi-structured interviews to determine the effect of embryo transfer timing on patient satisfaction/stress levels in participants who achieved a live birth and on closure/acceptance in those who did not get pregnant.
Incidence of facilitators and barriers for patient involvement | month 9 after embryo transfer
  The investigators will utilize a mixed-methods framework to identify facilitators and barriers for patient involvement in decision-making and implementation /dissemination of blastocyst embryo transfer in routine infertility care settings.

OTHER OUTCOMES:
cumulative live birth rate among participants with 1-2 vs 3-5 zygotes | month 9 after embryo transfer
  subgroup analysis of the cumulative live birth rate per egg retrieval in patients with very low (1-2) and higher number of embryos (3-5)
cumulative live birth rate among participants age <38 and ≥ 38 years | month 9 after embryo transfer
  subgroup analysis of the cumulative live birth rate per egg retrieval in patients <38 and ≥ 38 years

CONTACTS AND LOCATIONS:
Overall Officials: Werner Neuhausser, MD PhD, Principal Investigator — Beth Israel Deaconess Medical Center/Harvard Medical School; Dustin Rabideau, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Boston IVF, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No